CLINICAL TRIAL: NCT00735722
Title: A Prospective Randomized Trial Comparing Freedom From Atrial Fibrillation at One Year Post CABG in Patients Undergoing Concomitant Left Atrial Ablation Using HIFU Versus CABG in Patients With Persistent or Long Standing Persistent AF
Brief Title: A(f)MAZE-CABG Study
Acronym: AFMAZE-CABG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AF07004AF
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Coronary Arteriosclerosis; Atrial Fibrillation; Coronary Artery Bypass Graft Surgery
Keywords: AF; CAD
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concomitant HIFU ablation (Active Comparator): HIFU AF Ablation
  Interventions: Device: HIFU AF Ablation
- Best medical treatment (No Intervention): Best medical treatment

INTERVENTIONS:
Device: HIFU AF Ablation — Concomitant left atrial ablation using High Intensity Focused Ultrasound (HIFU)
  Other Names: • Epicor™ UltraCinch™ LP Ablation Device; • Epicor™ UltraWand™ LP Tissue Ablation Wand; • Epicor™ LP Positioning and Sizing (LP PAS™) System; • Epicor™ LP Oblique Introducer
  Arms: Concomitant HIFU ablation

SUMMARY:
Concomitant AF ablation with HIFU in patients with persistent or long standing persistent AF undergoing CABG will be superior in restoring SR, compared with patients with persistent or long standing persistent AF undergoing CABG treated with best medical treatment according to ACC/AHA/ESC 2006 guidelines and no AF ablation.

DETAILED DESCRIPTION:
Primary Objective

• To compare the efficacy of concomitant AF ablation using HIFU to no ablation at 12 months in patients with persistent or long standing persistent AF undergoing CABG according to ACC/AHA/ESC 2006 guidelines and HRS/EHRA/ECAS Consensus Statement on Catheter and Surgical Ablation .

Secondary Objectives

* To compare the safety of concomitant AF ablation using HIFU to no ablation in patients with persistent or long standing persistent AF undergoing CABG.
* To compare AF burden in patients with persistent or long standing persistent AF treated with concomitant HIFU AF ablation undergoing CABG to those receiving no ablation.
* To compare the quality of life of patients with persistent or long standing persistent AF treated with concomitant HIFU AF ablation undergoing CABG to those receiving no ablation.
* To compare the health economic impact of concomitant AF ablation with HIFU in patients with persistent or long standing persistent AF undergoing CABG to those receiving no ablation.
* To compare the morbidity associated with persistent or long standing persistent AF in patients following CABG and ablation compared to those receiving no ablation.
* To compare cardiac function and left atrial transport associated with persistent or long standing persistent AF patients following CABG and ablation compared to those receiving no ablation.
* To document the incidence of immediate post ablation bidirectional conduction block through the pulmonary venous cinch and mitral lines.
* To document the effect of Intra-operative pre and post ablation stimulation and ablation of the autonomic ganglia.

ELIGIBILITY:
Inclusion Criteria:

* Legal age in host country
* Scheduled for CABG surgery
* Patient suffering from persistent or long-standing persistent AF
* Patients having the ability to fully comply with the study requirements
* Life expectancy > 2 years
* Patients who have given written informed consent to participate in the study

Exclusion Criteria:

* Clinically significant local or systemic infection or active endocarditis
* Sutures, pacing/defibrillator leads on the left side of the heart, valve prostheses or rings, or other implanted material in or adjacent to target treatment area.
* Stent in the coronary artery preventing an adequate mitral line
* Any other concomitant operation on the heart
* Previous heart surgery
* Patients who are or may potentially be pregnant
* Previous catheter ablation for atrial arrhythmia
* LA size more than 60 mm in apical view on Trans-Thoracic Echocardiogram (TTE)
* LA thrombus on intra-operative Trans-Oesophageal Echocardiogram (TOE)
* Known contraindication to Amiodarone
* Inability to undergo TOE
* Patients who are unable to give full informed consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Freedom from Atrial Arrhythmias (AF, Atrial Flutter, Atrial Tachycardia) at 12 months | 12 months

SECONDARY OUTCOMES:
Freedom from AF and other atrial arrhythmias at 3, 6, 9 and 18 months post ablation procedure (determined by 24 hour Holter monitor) | 18 months
Freedom from AF and other atrial arrhythmias at 24 months post ablation procedure (determined by 72 hour Holter monitor) | 24 months
AF burden (determined by 24 and 72 hour Holter monitor). | 24 months
Morbidity performing concurrent ablation in patients undergoing CABG assessed using length of ICU and hospital stay | 24 months
Incidence of stroke, TIA, PV stenosis, bleeding, thromboembolic complications, subsequent pace maker implantation, and death | 24 months
LV function and dimensions and LA size/transport capability | 24 months
Incidence of conduction block post ablation both intraoperatively across the pulmonary venous and mitral lines | At intervention
Effect of autonomic ganglia stimulation pre and post ablation intra-operatively | Discharge
Quality of life measurements (SF-36) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Dalrymple-Hay, Mr., Principal Investigator — Derriford Hospital, Plymouth, United Kingdom
Locations (10):
- Canada (2):
  - Queen Elisabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- Tampere University Hospital, Tampere, Western Finland, Finland
- Germany (2):
  - Herzzentrum Essen, Essen, North Rhine-Westphalia
  - Universitatsklinikum Schleswig Holstein Campus Luebeck, Lübeck, Schleswig-Holstein
- Catharina Ziekenhuis, Eindhoven, North Brabant, Netherlands
- Norway (2):
  - Feiringklinikken, Feiring
  - Rikshospitalet, Oslo
- United Kingdom (2):
  - Derriford Hospital, Plymouth, Devon
  - Southampton University Hospital, Southampton, Hampshire